CLINICAL TRIAL: NCT01616498
Title: Obesity and Muscle Function Pilot Study
Brief Title: Lean Muscle Function
Acronym: LEAN
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Barbara Nicklas, PhD, Professor, Wake Forest University Health Sciences
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00019632
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Single Muscle Fibers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma to be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lean: Comparison data from this lean cohort will be compared to the obese older adults are already being collected in an R01-funded study (Improving Muscle for Functional Independence Trial; IRB00009098; NCT01049698)

SUMMARY:
This pilot study is designed to determine the relationship between intra-myocellular lipids and muscle contractility in fibers from obese and non-obese older adults. Obese participants are being recruited for an on-going weight loss intervention study and this application seeks approval to recruit and enroll a lean comparison group of non-obese older adults. The primary goal of this study is to characterize the contractile properties of single muscle fibers and whole muscle in healthy, non-obese individuals under the same recording conditions the investigators used for the obese population to begin to determine whether fat infiltration accounts for diminished force.

ELIGIBILITY:
Inclusion Criteria:

* Age=65-75 years
* BMI=18-24 kg/m2
* No resistance training for past 6 months
* Normal cognitive function (MMSE >24)
* No contraindications for participation in weight loss or weight lifting exercise including severe arthritis or musculoskeletal disorders, knee or hip replacement or spinal surgery in past year
* Able to provide own transportation to study visits
* Not involved in any other research study involving strength training or undergoing physical therapy
* Not dependent on a cane or walker
* Willing to provide informed consent

Exclusion Criteria:

* Weight loss or gain (±5%) in past 6 months
* Body mass >136 kg (DXA limit)
* Current smoker (No nicotine within past year) or evidence of alcohol or drug abuse
* Insulin dependent or uncontrolled diabetes (FBG >140 mg/dL)
* Uncontrolled hypertension (BP>180/100 mmHg)
* Abnormal kidney function or liver blood tests
* Serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>2 mm) on ECG
* Past or current cardiovascular disease, including uncontrolled angina or dysrhythmia, hypertrophic cardiomyopathy, congestive heart failure, PAD, stroke, history of myocardial infarction, use of defibrillator or major heart surgery, or deep vein thrombosis or pulmonary embolus. These will be reviewed on a case by case basis.
* Past or current respiratory disease (requiring steroid treatment or supplemental oxygen)
* Past or current clinical diagnoses of neurological or hematological disease
* Use of any medications that could influence study variables (growth/steroid hormones, prescription anti-inflammatory medications, or beta blockers, Coumadin or any other blood thinner, including Plavix, Ticid, and Aggrenox)
* Cancer requiring treatment in past 2 years, except non-melanoma skin cancers
* Clinically evident edema or anemia

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 20 sedentary, normal-weight (BMI= 18-24 kg/m2) older (65-75 yrs) men and women (n=10 each)
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Muscle Fiber | Baseline
  Primary Aim:
  To measure single muscle fiber contractile properties, including specific force, unloaded shortening velocity, and maximum power. We will also measure whole muscle strength and size and fiber fat infiltration. These results will establish a reference database against which data recorded in older obese individuals can be compared.
  Primary hypothesis: Single muscle fibers will exhibit more force and power in healthy non-obese than obese older adults due to greater intra-myocellular fat infiltration.

SECONDARY OUTCOMES:
Muscle Strength | Baseline
  Non-obese older adults will exhibit greater whole muscle strength (absolute and relative to muscle mass and volume) and power than obese, older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available upon email request to the study PI and upon completion of a data-sharing agreement. This agreement will require that data be used only for research purposes, that no attempts be made to identify individual patients, that the data will be kept secure, that the user will not distribute the data to other researchers, that the user will return the files or destroy them once the project is completed, and that the user will acknowledge the data source. All data files will be de-identified. In addition, variables that could permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects will be removed or recoded. We will create a link on our website that describes our study and the data available for data sharing with descriptions.